CLINICAL TRIAL: NCT04482842
Title: Gene-guided Warfarin for Anticoagulation Therapy in Patients With Acute Ischemic Stroke
Brief Title: Gene-guided Warfarin for Anticoagulation Therapy
Acronym: GWAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-067
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gene-guided Warfarin (Experimental)
  Interventions: Device: Gene detection (CYP2C9*3, VKORC1); Drug: Warfarin Sodium
- Routine use (Other)
  Interventions: Drug: Warfarin Sodium

INTERVENTIONS:
Device: Gene detection (CYP2C9*3, VKORC1) — Warfarin is administered at the recommended dose by detecting CYP2C9*3 and VKORC1 gene polymorphismsand. The doctor adjusts the dosage according to the fluctuation of INR value in time.
  Arms: Gene-guided Warfarin
Drug: Warfarin Sodium — Warfarin is administered at a gene-guided dose or at a regular dose.

SUMMARY:
This study will explore the effect of warfarin gene polymorphism on the effectiveness and safety of anticoagulant therapy in patients with acute ischemic stroke, and clarify the correlation between genetic testing and compliance rate of INR value. It will illustrate the significance of gene-guided warfarin for administered dose to anticoagulation therapy in patients with acute ischemic stroke. Then it will establish and verify a warfarin stable dose prediction model suitable for such patients, and provide basis for the personalized medication regimen of warfarin in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke aged ≥18 years (cardiogenic cerebral embolism patients)
* Clinicians judge that long-term oral anticoagulation with warfarin is required
* No anticoagulation treatment in the past 10 days
* Agree to participate in this project

Exclusion Criteria:

* Patients who had a tendency to bleed when taking warfarin
* High-risk groups using warfarin anticoagulation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Stroke recurrence rate, compliance rate of INR value | 12 months
  Evaluation and analysis of the stroke recurrence rate and compliance rate of INR value at 12 months after treatment

IPD SHARING:
Plan to Share IPD: Undecided